CLINICAL TRIAL: NCT06506357
Title: A Single Group Study to Evaluate the Effects of a Probiotic Supplement on Vaginal Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Love Wellness (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20433
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Vaginal Health; Women's Health
Keywords: Probiotic Supplement; Urinary Tract Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic Supplement Group (Experimental): Participants in this group will receive the Good Girl Probiotics supplement.
  Interventions: Dietary Supplement: Good Girl Probiotics

INTERVENTIONS:
Dietary Supplement: Good Girl Probiotics — Participants will take one capsule of the Good Girl Probiotics supplement daily in the morning for eight weeks.

SUMMARY:
This virtual single-group clinical trial aims to evaluate the effects of the Good Girl Probiotics supplement on vaginal health. Participants will take one capsule of the probiotic supplement daily for eight weeks. They will complete questionnaires at Baseline, after the first dose, and at the end of Weeks 2, 4, 6, and 8 to assess changes in vaginal pH, vaginal health, and urinary tract health.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth.
* Aged 18+.
* Interested in supporting a balanced vaginal pH, vaginal health, and urinary tract health.
* Regularly experience symptoms of an unbalanced vagina, including an atypical smell, discharge, itching, swelling, irritation, pain during sex, and/or burning sensation while urinating.
* Willing to avoid using products or medications that target vaginal or urinary tract health infections.
* Willing to avoid other probiotics.
* Able to follow the study protocol.

Exclusion Criteria:

* Two or more bladder infections in six months or three or more infections in a year.
* Recent surgeries or invasive treatments within the last six months.
* Use of products or medications targeting vaginal or urinary tract health in the last 12 weeks.
* Known allergies to the product ingredients.
* Chronic health conditions impacting participation.
* Pregnant, breastfeeding, or trying to conceive.
* History of substance abuse.
* Current or former smoker within the past six months.
* Participation in another clinical trial.
* Diagnosed vaginal or pelvic conditions.
* Use of vaginal-related birth control (NuvaRing, IUD).
* Changes in hormonal birth control in the last three months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Vaginal and Urinary Tract Health and Balance | Baseline, Week 2, Week 4, Week 6, Week 8
  Assessment of vaginal and urinary tract health and balance through questionnaires completed by participants at Baseline, after the first dose, and at the end of Weeks 2, 4, 6, and 8.

SECONDARY OUTCOMES:
Vaginal Environment and Odor | Baseline, Week 2, Week 4, Week 6, Week 8
  Assessment of the vaginal environment and odor through questionnaires completed by participants at Baseline, after the first dose, and at the end of Weeks 2, 4, 6, and 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No